CLINICAL TRIAL: NCT00464737
Title: A Parallel, Randomized, Double-Blind, Placebo-Controlled, Multicenter Proof of Concept Trial to Assess the Efficacy and Safety of 2 Different Doses of Rotigotine in Subjects With Signs and Symptoms Associated With Fibromyalgia Syndrome
Brief Title: The Use of Rotigotine for Treatment of Reducing Signs and Symptoms of Fibromyalgia in Adults.
Acronym: SP888
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP888
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2010-01-05 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2010-09

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndrome; Rotigotine; Neupro
MeSH Terms: conditions — Fibromyalgia | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Rotigotine 4 mg (Experimental): 4 mg/24 hrs
  Interventions: Drug: Rotigotine
- Rotigotine 8 mg (Experimental): 8 mg/24 hrs
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Titration by Week 4 to two 20 cm2 patches (one placebo patch and one 4 mg/24 hrs patch)
  Other Names: Neupro
  Arms: Rotigotine 4 mg
Drug: Rotigotine — Titration by Week 4 to two 20 cm2 patches (both are 4 mg/24 hrs patches)
  Other Names: Neupro
  Arms: Rotigotine 8 mg
Other: Placebo — Titration by Week 4 to two 20 cm2 placebo patches. At all weeks, placebo patches are matched in size and appearance to active patches.
  Arms: Placebo

SUMMARY:
This trial is to investigate the efficacy and safety of rotigotine as compared to placebo in reducing signs and symptoms of fibromyalgia syndrome. The effects of rotigotine on pain, sleep, general activity, mood, and quality of life, and the use of rescue medication to treat pain will be assessed.

DETAILED DESCRIPTION:
The overall post-Baseline duration of treatment was 13 weeks. The trial consisted of a 4-week Titration Phase, an 8-week Maintenance Phase, a 1-week De-escalation Phase, and a 2-week Safety Follow-Up Phase. If subjects met the eligibility criteria, they were randomized to receive rotigotine 4 mg/24 hrs, rotigotine 8 mg/24 hrs, or placebo during the Maintenance Phase. During the 4-week Titration Phase, subjects assigned to rotigotine were titrated at weekly intervals of 2 mg/24 hrs until they reached 4 mg/24 hrs or 8 mg/24 hrs. All subjects who completed the 4-week Titration Phase entered an 8-week Maintenance Phase and were maintained at their randomized dose (rotigotine 4 mg/24 hrs, rotigotine 8 mg/24 hrs, or placebo). No dose adjustment was allowed during the Maintenance Phase. The Treatment Phase was defined as the combined Titration and Maintenance Phases.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 18 to 65 years of age (inclusive)
* Subject fulfills all 3 points of the American College of Rheumatology (ACR) definition for diagnosis of fibromyalgia (pain, stiffness, and/or sleep disorder)
* Subject must complete an adequate washout period for excluded medications, as necessary, prior to beginning the Baseline Diary Phase
* Subject has at least moderate pain that is defined as an average pain intensity of ≥5 on an 11-point Likert pain scale (0-10) during the 7 days prior to Baseline
* Subject must have at least 5 morning and 5 evening Likert pain scale scores for the 7 days immediately prior to Visit 2 and the average daily pain score over these 7 days must be ≥5 (average daily pain score is determined as follows: calculate the mean of the morning and evening scores separately using all pain scores for the 7 days immediately prior to Visit 2; add the mean morning and evening scores and divide by 2)
* Subject has a score of ≥50 on Fibromyalgia Impact Questionnaire (FIQ), with a score of 100 representing severe disease at Baseline

Exclusion Criteria:

* Subject has symptomatic regional or structural rheumatic disease (eg, knee or hip osteoarthritis, bursitis, tendonitis), rheumatic autoimmune disease or inflammatory rheumatic disease, such as systemic lupus erythematosus (SLE), mild primary osteoarthritis of the hand(s) is allowed
* Subject has diagnosed neuropathic pain syndrome
* Subject has received therapy with a dopamine agonist (eg, pramipexole, ropinirole) for 3 months or longer that was not considered effective in managing fibromyalgia symptoms
* Subject is receiving disability or is involved in litigation related to fibromyalgia syndrome
* Subject has significant psychopathology as determined by the investigator based on results of the Structural Clinical Interview for DSM-IV Diagnosis (SCID-I). The SCID-I must be administered by a physician or clinical psychologist trained to administer the instrument
* Subject has evidence of an impulse control disorder according to the Jay Modified Minnesota Impulsive Disorders Interview (MIDI)
* Subject has any medical condition that, in the opinion of the investigator, could jeopardize or compromise the subject's ability to participate in this trial
* Subject has orthostatic hypotension with a decrease of blood pressure (BP) from supine to standing position of ≥20 mmHg in systolic blood pressure (SBP) or of ≥10 mmHg in diastolic blood pressure (DBP) taken from the 5-minute supine value and the 1- and/or 3-minute standing measurements, or supine SBP <105 mmHg at Baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (35):
- United States (35):
  - Mobile, Alabama
  - Mesa, Arizona
  - Peoria, Arizona
  - Santa Ana, California
  - Cromwell, Connecticut
  - DeLand, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Beach, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Columbia, Maryland
  - Springfield, Massachusetts
  - St Louis, Missouri
  - Stratford, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Rochester, New York
  - Williamsville, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Souderton, Pennsylvania
  - Crossville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Woodstock, Vermont
  - Richmond, Virginia
  - Seattle, Washington

REFERENCES:
- See also: For Safety Alerts amd Recalls refer to — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Full Analysis Set (FAS) contains all randomized subjects who received at least 1 dose of trial medication, and had at least 1 post-Baseline Likert pain score. The Per Protocol Set contains all subjects in the FAS who completed at least 2 weeks of the Maintenance Phase and had no major protocol deviations.
Pre-assignment Details: Participant flow is based on the 230 randomized subjects however 1 subject randomized to Rotigotine 4 mg/24 hrs did not receive study medication and was excluded from the Safety Set. Thus 229 subjects are included in summaries of baseline characteristics and adverse events. The excluded subject was a 47-year old female enrolled in the United States
Groups:
- Rotigotine 4 mg: Rotigotine 4 mg/24 hrs
- Rotigotine 8 mg: Rotigotine 8 mg/24 hrs
Period: Overall Study
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Started | 82 | 74 | 74
Completed | 50 | 42 | 19
Not Completed | 32 | 32 | 55
Not completed — Adverse Event | 12 | 17 | 33
Not completed — Lack of Efficacy | 7 | 7 | 4
Not completed — Withdrawal by Subject | 5 | 3 | 5
Not completed — Protocol Violation | 1 | 1 | 5
Not completed — Non-compliance | 0 | 1 | 1
Not completed — Lost to Follow-up | 5 | 2 | 5
Not completed — Other: Subject's schedule doesn't permit | 1 | 0 | 0
Not completed — Other: Subject left town; family illness | 1 | 0 | 0
Not completed — Other: Study demands too great | 0 | 1 | 0
Not completed — Other: Personal family reasons | 0 | 0 | 1
Not completed — Other: Subject's disability per sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg | Total
Number analyzed (Participants) | 82 | 73 | 74 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 81 | 73 | 73 | 227
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (10.7) | 47.5 (10.3) | 47.0 (11.6) | 47.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 65 | 68 | 209
  Male | 6 | 8 | 6 | 20
Region of Enrollment [Number; unit: participants]
  United States | 82 | 73 | 74 | 229

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Pain Score to the Last 2 Weeks of the 12-week Treatment Phase (Based on the Full Analysis Set)
Description: The average daily pain score is calculated using an 11-point Likert scale, ranging from 0 (no pain) to 10 (worst pain ever experienced).
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: Of the 82 (Placebo), 74 (Rotigotine 4 mg), and 74 (Rotigotine 8 mg) patients randomized, 81, 70 and 72 patients respectively are included in the summary of the last 2 weeks of the 12-week Treatment Phase, based on the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 81 | 70 | 72
Score on a scale | -1.12 (1.83) | -1.27 (1.86) | -0.83 (1.70)

2. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) Total Score to the Last Assessment in the 12-week Treatment Phase
Description: The Fibromyalgia Impact Questionnaire (FIQ) Total Score ranges from 0 to 100 with higher scores corresponding to a greater impact of fibromyalgia
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: Of the 82 (Placebo), 74 (Rotigotine 4 mg), and 74 (Rotigotine 8 mg) patients randomized, 80, 64 and 63 patients respectively are included in this summary based on the Full Analysis Set and have the Last Assessment in the 12-week Treatment Phase.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 80 | 64 | 63
Score on a scale | -14.9 (15.6) | -13.4 (13.7) | -12.8 (18.1)

3. Secondary Outcome: Change From Baseline in Total Myalgic Score to the Last Assessment in the 12-week Treatment Phase
Description: Total Myalgic Score ranges from 0 to 54 with higher scores corresponding to a greater level of pain.
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: Based on the observed outcome for the primary efficacy variable for this study, an abbreviated clinical study report was produced. Summaries were not produced for all pre-planned outcome measures and thus these results are not available. This summary was not produced for the abbreviated clinical study report.
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Average Daily Interference With Sleep to the Last 2 Weeks of the 12-week Treatment Phase
Description: Sleep scale - the subject rated quality of sleep, from 0 (very good sleep) to 10 (very poor sleep)
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 81 | 70 | 72
Score on a scale | -0.95 (2.01) | -0.82 (2.03) | -0.48 (2.09)

5. Secondary Outcome: Change From Baseline in Daily Interference With General Activity to the Last 2 Weeks of the 12-week Treatment Phase
Description: General activity scale - the subject rated how the pain had interfered with general activity, from 0 (did not interfere) to 10 (completely interfered)
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 81 | 70 | 72
Score on a scale | -1.11 (2.05) | -1.19 (1.82) | -0.88 (2.10)

6. Secondary Outcome: Patient Global Impression of Change (PGIC) Assessment From Baseline to the Last Assessment in the 12-week Treatment Phase
Description: The PGIC is a 7-point self-administered categorical rating scale in which the subject rated the change in pain since starting trial medication (from much worse [score of 1] to much better [score of 7]).
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: Of the 82 (Placebo), 74 (Rotigotine 4 mg), and 74 (Rotigotine 8 mg) patients randomized, 76, 58, and 51 patients respectively are included in this summary based on the Full Analysis Set and have the Last Assessment in the 12-week Treatment Phase.
Measure: Number; unit: Patients
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 76 | 58 | 51
Patients
  Much better | 8 | 10 | 9
  Moderately better | 14 | 14 | 7
  Mildly better | 25 | 12 | 11
  No change | 16 | 17 | 12
  Mildly worse | 5 | 3 | 5
  Moderately worse | 7 | 1 | 5
  Much worse | 1 | 1 | 2

7. Secondary Outcome: Change From Baseline in Morning and Evening Pain Scores to the Last 2 Weeks of the 12-week Treatment Phase
Description: An 11-point Likert scale was used for subjects to assess pain, from 0 (no pain) to 10 (worst pain ever experienced).
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 81 | 70 | 72
Score on a scale
  Morning Pain Score | -1.07 (1.91) | -1.30 (1.91) | -0.78 (1.78)
  Evening Pain Score | -1.17 (1.82) | -1.24 (1.90) | -0.88 (1.89)

8. Secondary Outcome: Number of Subjects Using Rescue Medication and Alcohol During the 12-week Treatment Phase
Description: Subjects recorded use of rescue medication for pain in the diary daily in the evening with a Yes/No response. Use of alcohol to treat pain in the past 24 hours was recorded with a Yes/No response.
Time Frame: 12-week Treatment Phase
Population: as for outcome 3
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Rotigotine Plasma Concentration at the End of the Maintenance Phase/Week 12
Time Frame: End of the Maintenance Phase/Week 12
Population: The number of patients in the Placebo group has been presented as 0 as this outcome measure is not applicable for this treatment group. Of the 73 (Rotigotine 4 mg) and 74 (Rotigotine 8 mg) patients respectively in the Safety Set, a total of 41 and 20 patients respectively at the end of Maintenance Phase/Week 12 have this assessment.
Measure: Mean (Standard Deviation); unit: ug/ML
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 0 | 41 | 20
ug/ML |  | 0.2388 (0.2337) | 0.2981 (0.2973)

10. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Scores to the Last Assessment in the 12-week Treatment Phase
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-administered instrument for detecting anxiety and depression in medical outpatients. Scores range from 0 to 21 for each subscale with higher scores reflecting a greater level of anxiety or depression.
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: as for outcome 3
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Fibromyalgia Symptom Scores to the Last Assessment in the 12-week Treatment Phase
Description: All scores range from 0 to 10 with higher scores corresponding to a greater level of symptom severity.
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: as for outcome 3
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II (BDI-II) Scores to the Last Assessment in the 12-week Treatment Phase
Description: The Beck Depression Inventory-II is a 21-item questionnaire. Each item is scored on a scale of 0 to 3 with a total score ranging from 0 to 63. A higher total score is associated with more severe depressive symptoms.
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: as for outcome 3
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With Presence of Impulse Control Disorders
Description: Impulse control disorders (ICDs) are a set of psychiatric disorders in which a person is unable to control strong and often harmful impulses. They are assessed in this study using the Jay Modified Minnesota Impulsive Disorders Interview (Jay Modified MIDI), which focuses on the five most common ICDs that may be associated with dopamine agonist use: compulsive buying, compulsive gambling, compulsive eating, hypersexuality and punding (performing repetitive and/or mechanical tasks).
Time Frame: 12-week Treatment Phase
Population: as for outcome 3
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 0 | 0 | 0

14. Primary Outcome: Change From Baseline in Average Daily Pain Score to the Last 2 Weeks of the 12-week Treatment Phase (Based on the Per Protocol Set)
Description: as for outcome 1
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: Of the 82 (Placebo), 74 (Rotigotine 4 mg), and 74 (Rotigotine 8 mg) patients randomized, 50, 33 and 22 patients respectively are included in the summary of the last 2 weeks of the 12-week Treatment Phase, based on the Per Protocol Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Number analyzed (Participants) | 50 | 33 | 22
score on a scale | -1.28 (1.79) | -2.09 (2.07) | -1.57 (2.27)

ADVERSE EVENTS:
Description: The Safety Set (SS) is comprised of all subjects who received at least 1 dose of trial medication.
Arm/Group | Placebo | Rotigotine 4 mg | Rotigotine 8 mg
Serious Adverse Events (participants affected / at risk) | 4/82 | 1/73 | 1/74
Other Adverse Events (participants affected / at risk) | 53/82 | 55/73 | 65/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Rotigotine 4 mg (N=73) | Rotigotine 8 mg (N=74)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Rotigotine 4 mg (N=73) | Rotigotine 8 mg (N=74)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (6) | 5 (5) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 5 (5) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 5 (6) | 7 (7)
Nausea (Gastrointestinal disorders) | 18 (25) | 34 (46) | 48 (63)
Vomiting (Gastrointestinal disorders) | 1 (1) | 13 (15) | 18 (22)
Application site irritation (General disorders) | 1 (1) | 6 (6) | 5 (6)
Application site pruritus (General disorders) | 4 (5) | 3 (3) | 11 (11)
Fatigue (General disorders) | 2 (4) | 5 (6) | 1 (1)
Sinusitis (Infections and infestations) | 6 (7) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 7 (7) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 6 (6) | 10 (10) | 8 (10)
Headache (Nervous system disorders) | 12 (17) | 13 (18) | 12 (15)
Somnolence (Nervous system disorders) | 6 (6) | 8 (9) | 7 (9)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (10) | 7 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.